CLINICAL TRIAL: NCT02417844
Title: Single Center, Single Dose, Open-label, Randomized, Two-way Crossover Study to Determine Bioequivalence of Two Formulations Containing Tamsulosin HCl 04.mg MR Capsules in at Least 30 Healthy Male Subjects Under Fed Conditions
Brief Title: Determine the Bioequivalence of Two Formulations of Tamsulosin HCl Capsules in Fed Male.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 527.89
Record Dates: First submitted 2015-04-13; First posted 2015-04-16 (Estimated); Results first posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tamsulosin

ARMS (2):
- Tamsulosin HCl (Active Comparator)
  Interventions: Drug: Tamsulosin HCL
- Tamsulosin (Active Comparator)
  Interventions: Drug: tamsulosin (Astellas)

INTERVENTIONS:
Drug: tamsulosin (Astellas)
  Arms: Tamsulosin
Drug: Tamsulosin HCL
  Arms: Tamsulosin HCl

SUMMARY:
Two tamsulosin HClformulations will be tested in fed state

ELIGIBILITY:
Inclusion criteria:

Health male volunteers 18 years and older

Exclusion criteria:

History of hypersensitivity or allergy to IMP or its excipients or any related medication

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2015-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each treatment was administered after consumption of a high-fat, high-calorie breakfast.
Groups:
- Tamsulosin HCl (Test) / Flomax Relief (Reference): Oral administration of Tamsulosin hydrochloride (HCl) 0.4mg modified release (MR) capsule followed by oral administration of Flomax Relief modified release (MR) 0.4mg capsule (tamsulosin MR capsules).
- Flomax Relief (Reference) / Tamsulosin HCl (Test): Oral administration of Flomax Relief modified release (MR) 0.4mg capsule (tamsulosin MR capsules) followed by oral administration of Tamsulosin hydrochloride (HCl) 0.4mg modified release (MR) capsule.
Period: Overall Study
Arm/Group | Tamsulosin HCl (Test) / Flomax Relief (Reference) | Flomax Relief (Reference) / Tamsulosin HCl (Test)
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set which included all subjects who received at least one dose of investigational medicinal product.
Groups:
- All Subjects: Subjects each received two treatments which were each administered orally and separated by a washout period of 7 days. The treatments were:
  * Flomax Relief (Reference): Flomax Relief modified release (MR) 0.4mg capsule (tamsulosin MR capsules).
  * Tamsulosin hydrochloride (HCl) (Test): Tamsulosin HCl 0.4mg modified release (MR) capsule.
Arm/Group | All Subjects
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24.6 (5.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 34

OUTCOME MEASURES:

1. Primary Outcome: Maximum Measured Concentration (Cmax)
Description: Maximum measured concentration of analyte in plasma (Cmax)
Time Frame: Before drug administration (0 hours (h)) and 1h, 2h, 3h, 4h, 5h, 6h, 6.5h, 7h, 7.5h, 8h, 10h, 12h, 16h, 24h, 36h, 48h and 72h after drug administration
Population: Pharmacokinetic (PK) set which included all subjects who had evaluable PK data for both treatment periods.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Groups:
- Tamsulosin HCl (Test): Oral administration of Tamsulosin hydrochloride (HCl) 0.4mg modified release (MR) capsule.
- Flomax Relief (Reference): Oral administration of Flomax Relief modified release (MR) 0.4mg capsule (tamsulosin MR capsule).
Arm/Group | Tamsulosin HCl (Test) | Flomax Relief (Reference)
Number analyzed (Participants) | 34 | 34
pg/mL | 8826 (31.8) | 8856 (34.0)
Statistical Analysis 1: Comparison: Tamsulosin HCl (Test) vs Flomax Relief (Reference); Test type: Non-Inferiority or Equivalence — Bioequivalence range of 80% to 125%; Geometric mean ratio (%) = 99.66, 90% CI 2-sided [92.19 to 107.74], Standard Deviation 19.15 — The standard deviation in the statistical analysis is actually the intra-individual coefficient of variation. Ratio calculated as test divided by reference

2. Primary Outcome: Area Under the Concentration-time Curve From 0 to the Time of the Last Quantifiable Concentration (AUC0-tz)
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable concentration (AUC0-tz)
Time Frame: as for outcome 1
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Tamsulosin HCl (Test) | Flomax Relief (Reference)
Number analyzed (Participants) | 34 | 34
h*pg/mL | 164700 (42.4) | 165400 (43.7)
Statistical Analysis 1: Comparison: Tamsulosin HCl (Test) vs Flomax Relief (Reference); Test type: Non-Inferiority or Equivalence — Bioequivalence range of 80% to 125%; Geometric mean ratio (%) = 99.58, 90% CI 2-sided [94.23 to 105.24], Standard Deviation 13.51 — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Area Under the Concentration-time Curve From 0 Extrapolated to Infinity (AUC0-inf)
Description: Area under the concentration-time curve of analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-inf).
Time Frame: as for outcome 1
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Tamsulosin HCl (Test) | Flomax Relief (Reference)
Number analyzed (Participants) | 34 | 34
h*pg/mL | 170100 (44.1) | 171000 (45.2)
Statistical Analysis 1: Comparison: Tamsulosin HCl (Test) vs Flomax Relief (Reference); Test type: Non-Inferiority or Equivalence — Bioequivalence range of 80% to 125%; Geometric mean ratio (%) = 99.48, 90% CI 2-sided [93.90 to 105.39], Standard Deviation 14.12 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax)
Description: Time from last dosing to the maximum plasma concentration (tmax).
Time Frame: as for outcome 1
Population: PK set
Measure: Median (Full Range); unit: Hours
Arm/Group | Tamsulosin HCl (Test) | Flomax Relief (Reference)
Number analyzed (Participants) | 34 | 34
Hours | 7.51 [4.00 to 12.01] | 8.00 [4.00 to 24.01]

5. Secondary Outcome: Terminal Elimination Rate Constant (λz)
Description: Terminal elimination rate constant in plasma (λz)
Time Frame: as for outcome 1
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Tamsulosin HCl (Test) | Flomax Relief (Reference)
Number analyzed (Participants) | 34 | 34
1/hour | 0.05 (21.6) [0.03 to 0.08] | 0.05 (21.9) [0.04 to 0.10]

6. Secondary Outcome: Apparent Terminal Elimination Half-life (t1/2)
Description: Apparent terminal elimination half-life of the analyte in plasma (t1/2)
Time Frame: as for outcome 1
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Tamsulosin HCl (Test) | Flomax Relief (Reference)
Number analyzed (Participants) | 34 | 34
hours | 13.16 (21.6) [9.12 to 20.10] | 13.21 (21.9) [6.93 to 18.70]

ADVERSE EVENTS:
Time Frame: Up to 72 hours
Groups:
- Flomax Relief (Reference): Oral administration of Flomax Relief modified release (MR) 0.4mg capsule (tamsulosin MR capsules).
Arm/Group | Tamsulosin HCl (Test) | Flomax Relief (Reference)
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 5/34 | 1/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tamsulosin HCl (Test) (N=34) | Flomax Relief (Reference) (N=34)
Headache (Nervous system disorders) | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.